CLINICAL TRIAL: NCT06466850
Title: The Efficacy of Allogenic Mesenchymal Stem Cells Derived Exosomes in Osteoarthritis Patients
Brief Title: Mesenchymal Stem Cells Derived Exosomes in Osteoarthritis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Dehghani, Dr, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Isfahan med
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Patients with moderate to severe osteoarthritis, Kellgren-Lawrence grade 2,3 in both knees; accompanied by mild to moderate pain and swelling are included.
  Interventions: Biological: Exosome

INTERVENTIONS:
Biological: Exosome — intra-articular injection is suggested for two times: day 1and day 90
  Other Names: EVs

SUMMARY:
Present research focuses on the potential of exosomes, which are small vesicles secreted by mesenchymal stem cells (MSCs), as a therapeutic approach for osteoarthritis (OA).

OA is a degenerative joint disorder characterized by the destruction of cartilage and loss of extracellular matrix. It's associated with pro-inflammatory cytokines and increased expression of matrix metalloproteinase (MMP) and "a disintegrin and metalloproteinase with thrombospondin motifs" (ADAMTS).

MSCs have been explored as a new treatment for OA over the last decade1. It's suggested that the paracrine secretion of trophic factors, in which exosomes play a crucial role, contributes to the mechanism of MSC-based treatment of OA.

Exosomes derived from MSCs may suppress OA development. They carry bioactive molecules of the parental cells, including non-coding RNAs (ncRNAs) and proteins and anti-inflammatory factors. These exosomes have shown a significant impact on the modulation of various physiological behaviors of cells in the joint cavity.

This research provides hope for developing more effective and predictable methods of using MSC-derived exosomes for OA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic history (for at least 3 months) of knee joint pain
* Body mass index (BMI) between 21.5 and 29.5
* Radiographically documented knee osteoarthritis of grades 1 to 3 (Kellgren-Lawrence (K-L) radiographic classification scale)

Exclusion Criteria:

* Rheumatoid arthritis and other rheumatic diseases
* Varus or valgus more than 10 degrees; lateral subluxation of the patella
* Deformity at the joint levels or adjacent to the knee due to fracture or any other injury
* Complete rupture of the ligament and meniscus leading to laxity or locking
* Serious systemic, oncohematological, autoimmune diseases; history of severe allergy; serious failure of vital organs, inability to walk
* Hyaluronic acid infiltration within the previous six months
* Hemoglobin levels <10 g/dL;

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis index (WOMAC) | 1, 3, and 6 months. The second injection is repeated in day 90 after first injection.
  Filling out the WOMAC questionnaire, evaluating the measures related to knee function

CONTACTS AND LOCATIONS:
Overall Officials: Leila Dehghani, Dr, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Leila Dehghani, Isfahan, Iran